CLINICAL TRIAL: NCT01196741
Title: A Randomised Placebo-controlled Trial of Saracatinib (AZD0530) Plus Weekly Paclitaxel in Platinum Resistant Ovarian, Fallopian Tube or Primary Peritoneal Cancer
Brief Title: Saracatinib and Paclitaxel in Platinum-resistant Ovarian Cancer
Acronym: SaPPrOC
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University College, London (Other)
Collaborators: AstraZeneca (Industry); Cancer Research UK (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: UCL/09/105; Funder reference (academic) (Other Grant/Funding Number: CRUK/10/007); Funder reference (industry) (Other Grant/Funding Number: ISS05300017); 2009-017171-13 (EudraCT Number)
Record Dates: First submitted 2010-09-01; First posted 2010-09-08 (Estimated); Results first posted 2015-05-05 (Estimated); Last update posted 2015-05-05 (Estimated); Status verified 2014-01

CONDITIONS: Ovarian Cancer; Fallopian Tube Cancer; Primary Peritoneal Cancer
MeSH Terms: conditions — Ovarian Neoplasms; Fallopian Tube Neoplasms | interventions — Paclitaxel; saracatinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Saracatinib plus weekly paclitaxel (Active Comparator)
  Interventions: Drug: Paclitaxel; Drug: Saracatinib
- Placebo plus weekly paclitaxel (Placebo Comparator)
  Interventions: Drug: Paclitaxel; Drug: Matched placebo

INTERVENTIONS:
Drug: Paclitaxel — Paclitaxel 80 mg/m2 weekly for 6 weeks followed by a 2 week break (1 cycle), for 4 cycles initially (32 weeks). If there is evidence of on-going response after 4 cycles, 3 further cycles will be given, unless there is dose-limiting toxicity or the patient requests to discontinue treatment. If best response is stable disease after 4 cycles, treatment should be discontinued but may continue at the discretion of the Investigator.
Drug: Saracatinib — Saracatinib 175 mg PO once daily, to begin 1 week prior to commencement of chemotherapy, taken continuously until progression
  Arms: Saracatinib plus weekly paclitaxel
Drug: Matched placebo — Matched placebo PO once daily, to begin 1 week prior to commencement of chemotherapy, taken continuously until progression
  Arms: Placebo plus weekly paclitaxel

SUMMARY:
The purpose of this study is to investigate whether the addition of the Src inhibitor saracatinib (AZD0530) to weekly paclitaxel improves efficacy, compared with paclitaxel plus placebo, in patients with relapsed platinum-resistant ovarian cancer. The trial will also determine toxicity and ascertain whether the combination of paclitaxel plus saracatinib should proceed to a phase III trial.

DETAILED DESCRIPTION:
A multicentre, randomised, double-blind, placebo-controlled Phase II trial will be conducted. The overall aim of the trial is to investigate whether the addition of saracatinib to weekly paclitaxel improves efficacy, as measured by progression free survival, compared with paclitaxel plus placebo. The trial will also determine toxicity and ascertain whether the combination of paclitaxel plus saracatinib should proceed to a phase III trial.

The toxicity data from Study NCT00610714 (D8180C00015) suggests that a small number of patients could experience febrile neutropaenia during their first chemotherapy cycle. To combat this, saracatinib (175 mg OD)/matched placebo will begin 1 week prior to commencement of chemotherapy, and be given continuously until progression.

All patients will receive cycles of weekly paclitaxel chemotherapy. One cycle will consist of weekly paclitaxel (80 mg/m2) for 6 weeks followed by 2 weeks rest. If there is evidence of on-going response after 4 cycles, 3 further cycles of saracatinib/placebo plus weekly paclitaxel will be given, unless there is dose-limiting toxicity or the patient requests to discontinue treatment. If best response is stable disease after 4 cycles, treatment should be discontinued but may continue at the discretion of the Investigator.

ELIGIBILITY:
Inclusion criteria:

* Confirmed relapsed ovarian, fallopian tube or primary peritoneal cancer AND relapse within the platinum-resistant (progression must not be based on Cancer Antigen 125 (CA125) alone) time-frame, i.e. have progressed within 6 months of platinum therapy.
* Patients need not have received prior taxane; if patients have received prior taxane, the interval since treatment must be known. Patients will be stratified as <6 months or 6+ months taxane interval/no prior taxane.
* Patients will generally have received at least 2 lines of prior chemotherapy, but may enter if they have relapsed within 6 months of first line therapy. Patients may have received prior liposomal doxorubicin, although this is NOT a requirement. The treatment immediately prior to study entry need not be platinum-based.
* Measurable or evaluable disease (if not measurable by Response Evaluation Criteria In Solid Tumours (RECIST) v1.1 criteria, patients must be evaluable by Gynecologic Cancer InterGroup (GCIG) CA125 criteria).
* Eastern Cooperative Oncology Group Performance Status (ECOG PS) 0-2
* Adequate haematological and biochemical function.

Exclusion criteria

* Prior administration of weekly paclitaxel.
* Tumours of malignant mixed mesodermal (MMMT) or mucinous subtypes, or non-epithelial ovarian cancers (e.g. Brenner tumours, Sex-cord tumours).
* Unresolved bowel obstruction.
* Chemotherapy within the preceding 3 weeks.
* Radiotherapy within the preceding 3 weeks.
* Treatment with any investigational agent within the preceding 4 weeks or within 5 half-lives of the investigational agent, whichever is longer.
* Known leptomeningeal involvement or intracranial disease.
* Evidence of interstitial lung disease (bilateral, diffuse, parenchymal lung disease).
* Resting ECG with measurable QTc interval of >480 msec at 2 or more time points within a 24 hour period.
* Pregnant or lactating females.
* Fertile women of childbearing potential not willing to use highly effective contraception for the duration of trial treatment and for at least 6 months after the last administration of saracatinib +/- paclitaxel.
* Inability or unwillingness to give informed consent.
* Ongoing active infection or a documented history of HIV infection, Hepatitis B or C.
* Concurrent congestive heart failure or prior history of New York Heart Association (NYHA) class III/IV cardiac disease.
* Concurrent autoimmune disorder, e.g. systemic lupus or any demyelinating disease.
* Use of immunosuppressive therapy or corticosteroids taken within the 4 weeks prior to study entry and during the treatment period.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2011-03; Primary Completion 2012-11 (Actual); Study Completion 2014-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Iain McNeish, Principal Investigator — Barts and the London NHS Trust
Locations (12):
- United Kingdom (12):
  - Addenbrooke's Hospital, Cambridge, Cambridgeshire
  - St Bartholomew's Hospital, London, Greater London
  - University College London Hospital, London, Greater London
  - Guy's Hospital, London, Greater London
  - The Royal Mardsen Hospital, London, Greater London
  - The Christie NHS Foundation Trust, Manchester, Greater Manchester
  - Mount Vernon Hospital, Rickmansworth, Middlesex
  - The Churchill Hospital, Oxford, Oxfordshire
  - Queen's Hospital, Burton-on-Trent, Staffordshire
  - Royal Marsden Hospital, Sutton, Surrey
  - St James's University Hospital, Leeds, Yorkshire
  - Beatson West of Scotland Cancer Centre, Glasgow

REFERENCES:
- [Derived] McNeish IA, Ledermann JA, Webber L, James L, Kaye SB, Hall M, Hall G, Clamp A, Earl H, Banerjee S, Kristeleit R, Raja F, Feeney A, Lawrence C, Dawson-Athey L, Persic M, Khan I. A randomised, placebo-controlled trial of weekly paclitaxel and saracatinib (AZD0530) in platinum-resistant ovarian, fallopian tube or primary peritoneal cancerdagger. Ann Oncol. 2014 Oct;25(10):1988-1995. doi: 10.1093/annonc/mdu363. Epub 2014 Jul 28. PMID 25070546

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Saracatinib Plus Weekly Paclitaxel | Placebo Plus Weekly Paclitaxel
Started | 71 | 36
Completed | 11 | 8
Not Completed | 60 | 28
Not completed — Disease progression | 34 | 14
Not completed — Adverse Event | 10 | 6
Not completed — Serious Adverse Event | 3 | 1
Not completed — Dose limiting Adverse Event | 2 | 1
Not completed — Withdrawal by Subject | 3 | 0
Not completed — Other reason | 3 | 3
Not completed — Other | 3 | 2
Not completed — Protocol Violation | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Saracatinib Plus Weekly Paclitaxel | Placebo Plus Weekly Paclitaxel | Total
Number analyzed (Participants) | 71 | 36 | 107
Age, Continuous [Median (Full Range); unit: years] | 62.8 [34.5 to 78.8] | 66.9 [20.0 to 82.1] | 63.4 [20.0 to 82.1]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 71 | 36 | 107
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United Kingdom | 71 | 36 | 107
Cancer Antigen 125 (CA125) [Median (Full Range); unit: U/mL] | 628 [8 to 12945] | 667 [24 to 7758] | 648 [8 to 12945]
Eastern Cooperative Oncology Group Performance Status (ECOG PS) [Number; unit: participants] — ECOG PS 0 = Fully active, able to carry out all normal (pre-disease) activity without restriction
  ECOG PS 1 = Restricted in physically strenuous activity but ambulatory and able to carry out light work, e.g. light house work, office work
  ECOG PS 2 = Ambulatory and capable of all self-care but unable to carry out any work activities. Up and about more than 50% of waking hours
  participants
    0 | 23 | 15 | 38
    1 | 45 | 20 | 65
    2 | 3 | 1 | 4
International Federation of Gynecology and Obstetrics(FIGO) Ovarian Cancer Staging at diagnosis [Number; unit: participants] — STAGE I: Tumour confined to ovaries
  STAGE II: Tumour involves one or both ovaries with pelvic extension (below the pelvic brim) or primary peritoneal cancer
  STAGE III: Tumour involves one or both ovaries with cytologically or histologically confirmed spread to the peritoneum outside the pelvis and/or metastasis to the retroperitoneal lymph nodes
  STAGE IV: Distant metastasis excluding peritoneal metastasis
  participants
    I | 6 | 2 | 8
    II | 5 | 1 | 6
    III | 45 | 31 | 76
    IV | 11 | 1 | 12
    Unknown | 4 | 1 | 5
Histological subtype [Number; unit: participants]
  High grade serous | 46 | 27 | 73
  Low grade serous | 4 | 2 | 6
  Clear cell | 6 | 1 | 7
  Grade 3 endometrioid | 2 | 2 | 4
  Grade 1/2 endometrioid | 3 | 1 | 4
  Undifferentiated | 7 | 2 | 9
  Unknown | 3 | 1 | 4
Prior Surgery [Number; unit: participants]
  Yes | 67 | 31 | 98
  No | 2 | 5 | 7
  Unknown | 2 | 0 | 2
Prior Taxane Interval [Number; unit: participants]
  <6 months | 15 | 8 | 23
  >=6 months/None | 56 | 28 | 84
Number of lines of Prior Chemotherapy [Number; unit: participants]
  1-2 | 43 | 19 | 62
  >2 | 26 | 17 | 43
  Unknown | 2 | 0 | 2
Number of lines of Prior Chemotherapy [Median (Full Range); unit: lines of chemotherapy] | 2.0 [1.0 to 7.0] | 2.0 [1.0 to 6.0] | 2.0 [1.0 to 7.0]

OUTCOME MEASURES:

1. Primary Outcome: 6 Month Progression-free Survival Rate (PFS) (Based on Combined Response Evaluation Criteria In Solid Tumours (RECIST) v1.1 +/- Gynecologic Cancer Intergroup (GCIG) CA125 Criteria)
Description: Where a patient's disease is not measurable by RECIST v1.1, response may be based on GCIG CA125 criteria plus symptoms.
  The 6 month progression-free survival rate will be calculated by the trial statistician during the final analysis.
Time Frame: Using RECIST v1.1 at baseline; at Week 7 or 8 of each chemotherapy cycle; and 3 monthly during follow up. CA125 response will be assessed at baseline, weeks 1, 3 and 6 of each chemotherapy cycle, and at every follow up visit.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Saracatinib Plus Weekly Paclitaxel | Placebo Plus Weekly Paclitaxel
Number analyzed (Participants) | 69 | 35
percentage of participants | 29 [22 to 37] | 34 [23 to 46]
Statistical Analysis 1: Comparison: Saracatinib Plus Weekly Paclitaxel vs Placebo Plus Weekly Paclitaxel; Test type: Superiority or Other; p = 0.57, Regression, Cox; Hazard Ratio (HR) = 0.89, 95% CI 2-sided [0.65 to 1.23]

2. Secondary Outcome: Overall Survival
Time Frame: First saracatinib/placebo dose until death, assessed up to 36 months
Measure: Median (Full Range); unit: months
Arm/Group | Saracatinib Plus Weekly Paclitaxel | Placebo Plus Weekly Paclitaxel
Number analyzed (Participants) | 69 | 35
months | 10.1 [8.3 to 16.2] | 12.3 [11.0 to 14.4]
Statistical Analysis 1: Comparison: Saracatinib Plus Weekly Paclitaxel vs Placebo Plus Weekly Paclitaxel; Test type: Superiority or Other; p = 0.81, Regression, Cox

3. Secondary Outcome: Objective Response Rate Based on Investigator Assessment Based on RECIST v1.1 +/- GCIG CA125 Criteria
Description: Where a patient's disease is not measurable by RECIST v1.1, response may be based on GCIG CA125 criteria plus symptoms.
Time Frame: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Saracatinib Plus Weekly Paclitaxel | Placebo Plus Weekly Paclitaxel
Number analyzed (Participants) | 69 | 35
percentage of participants | 29 | 43

4. Secondary Outcome: Median Duration of Response
Description: Where a patient's disease is not measurable by RECIST v1.1, response may be based on GCIG CA125 criteria plus symptoms.
  Duration of Response will be calculated by the trial statistician during the final analysis.
Time Frame: as for outcome 1
Reporting Status: Not Posted

5. Secondary Outcome: Quality of Life: Trial Outcome Index (TOI) Based on FACT-O
Description: The TOI value for each patient is derived at each timepoint by calculating the sum of 3 subscales: Physical Well-Being (PWB), Functional Well-Being (FWB), Additional Concerns. Each subscale score is derived from questions with 4 answers (0=not at all, 1=a little bit, 2=somewhat, 3=quite a bit, 4=very much). In each subscale reversals are performed and the individual question scores added together. This value is then multiplied by the number of questions within the subscale, and divided by the number of questions answered to derive a subscale score. The higher each subscale score, the better the QoL.
  PWB 7 questions, lower values=better QoL.
  FWB 7 questions, higher values=better QoL.
  Additional concerns 11 questions (higher values in 6 questions=better QoL; higher values in 5 questions=worse QoL)
  The TOI is reported for each arm based on the average TOI score of each patient calculated across the outcome measure time frame. The higher the TOI, the better the QoL.
Time Frame: Patients will fill in FACT-O questionnaires at the following timepoints: baseline; Weeks 1, 3 and 6 of every chemotherapy cycle; at every follow up visit
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Saracatinib Plus Weekly Paclitaxel | Placebo Plus Weekly Paclitaxel
Number analyzed (Participants) | 69 | 35
units on a scale | 66.89 (1.89) | 73.10 (2.56)
Statistical Analysis 1: Comparison: Saracatinib Plus Weekly Paclitaxel vs Placebo Plus Weekly Paclitaxel; Test type: Superiority or Other; p = 0.0476, Mixed Models Analysis

6. Secondary Outcome: Median Time To Progression Based on RECIST v1.1 and GCIG CA125 Criteria
Description: Where a patient's disease is not measurable by RECIST v1.1, response may be based on GCIG CA125 criteria plus symptoms.
  Time To Progression will be calculated by the trial statistician during the final analysis.
Time Frame: as for outcome 1
Reporting Status: Not Posted

7. Secondary Outcome: Median PFS
Time Frame: From first saracatinib/placebo dose to first documented progression and/or death, assessed up to 36 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Saracatinib Plus Weekly Paclitaxel | Placebo Plus Weekly Paclitaxel
Number analyzed (Participants) | 69 | 35
months | 4.7 [3.6 to 5.5] | 5.3 [3.6 to 7.2]
Statistical Analysis 1: Comparison: Saracatinib Plus Weekly Paclitaxel vs Placebo Plus Weekly Paclitaxel; Test type: Superiority or Other; p = 0.99, Regression, Cox

ADVERSE EVENTS:
Time Frame: From trial consent to 30 days after last administration of saracatinib/placebo.
Description: According to Common Terminology Criteria for Adverse Events (CTCAE) v4.0
Arm/Group | Saracatinib Plus Weekly Paclitaxel | Placebo Plus Weekly Paclitaxel
Serious Adverse Events (participants affected / at risk) | 40/69 | 18/35
Other Adverse Events (participants affected / at risk) | 20/69 | 7/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Saracatinib Plus Weekly Paclitaxel (N=69) | Placebo Plus Weekly Paclitaxel (N=35)
Anemia (Blood and lymphatic system disorders) | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 3 | 0
Neutrophil count decreased (Investigations) | 2 | 0
Vomiting (Gastrointestinal disorders) | 4 | 3
Abdominal pain (Gastrointestinal disorders) | 4 | 0
Diarrhea (Gastrointestinal disorders) | 3 | 2
Fever (General disorders) | 3 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 3 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Catheter related infection (Infections and infestations) | 0 | 1
Fatigue (General disorders) | 2 | 1
Abdominal distension (Gastrointestinal disorders) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 2 | 0
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 | 1
Skin infection (Infections and infestations) | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 1
Urinary tract infection (Infections and infestations) | 1 | 1
Anorexia (Metabolism and nutrition disorders) | 1 | 0
Ventricular arrthymia (Cardiac disorders) | 0 | 1
Creatinine increased (Investigations) | 1 | 0
Endocarditis infective (Infections and infestations) | 1 | 0
Fungal chest infection (Infections and infestations) | 1 | 0
Lung infection (Infections and infestations) | 1 | 0
Myocardial infarction (Cardiac disorders) | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Saracatinib Plus Weekly Paclitaxel (N=69) | Placebo Plus Weekly Paclitaxel (N=35)
Febrile neutropenia (Blood and lymphatic system disorders) | 3 | 0
Vomiting (Gastrointestinal disorders) | 4 | 3
Abdominal pain (Gastrointestinal disorders) | 4 | 0
Diarrhea (Gastrointestinal disorders) | 3 | 2
Fever (General disorders) | 3 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 3 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Participating sites may not publish trial results without prior written consent from the Trial Management Group